CLINICAL TRIAL: NCT06889987
Title: Efficacy of Bilateral Ultrasound Guided Intramuscular Quadratus Lumborum Plane Block (Ql4) Versus Bilateral Lateral Quadratus Lumborum Plane Block (Ql1) in Controlling Post-Operative Pain in Cancer Patient Undergoing Open Nephrectomy: A Randomized Control Study
Brief Title: Bilateral Ultrasound Guided Intramuscular Quadratus Lumborum Plane Block Versus Bilateral Lateral Quadratus Lumborum Plane Block in Controlling Postoperative Pain in Cancer Patients Undergoing Open Nephrectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Ahmed Ismail, Assistant Lecturer of Anesthesia, Pain Relief, and Intensive Care Unit, Faculty of Medicine, National Cancer Institute, Cairo University, Egypt., National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AP2412-201-088-194
Record Dates: First submitted 2025-03-16; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Bilateral; Ultrasound; Intramuscular Quadratus Lumborum Plane Block; Lateral Quadratus Lumborum Plane Block; Postoperative Pain; Cancer Patients; Open Nephrectomy
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthesia, General

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intramuscular quadratus lumborum group (Experimental): Patients will receive bilateral ultrasound-guided intramuscular quadratus lumborum block with an injection of 0.4 ml/kg bupivacaine 0.25% after induction of general anesthesia.
  Interventions: Drug: Intramuscular quadratus lumborum block
- Lateral quadratus lumborum group (Experimental): Patients will receive bilateral Ultrasound-guided lateral quadratus lumborum with injection of 0.4 ml/kg of bupivacaine 0.25 after induction of general anesthesia.
  Interventions: Drug: Lateral quadratus lumborum block
- Control group (Active Comparator): Patients will receive only general anesthesia without any block
  Interventions: Drug: General anesthesia

INTERVENTIONS:
Drug: Intramuscular quadratus lumborum block — Patients will receive bilateral ultrasound-guided intramuscular quadratus lumborum block with an injection of 0.4 ml/kg bupivacaine 0.25% after induction of general anesthesia
  Other Names: Bupivacaine 0.25%
  Arms: Intramuscular quadratus lumborum group
Drug: Lateral quadratus lumborum block — Patients will receive bilateral ultrasound-guided lateral quadratus lumborum with an injection of 0.4 ml/kg of bupivacaine 0.25 after induction of general anesthesia.
  Other Names: Bupivacaine 0.25%
  Arms: Lateral quadratus lumborum group
Drug: General anesthesia — Patients will receive only general anesthesia without any block.
  Arms: Control group

SUMMARY:
This study aims to evaluate the efficacy of bilateral ultrasound-guided intramuscular quadratus lumborum plane block (QL4) versus bilateral lateral quadratus lumborum plane block (QL1) in controlling postoperative pain in cancer patients undergoing open nephrectomy.

DETAILED DESCRIPTION:
Post-surgical somatic pain is very distressing to patients, which may lead to significant complications.

Practitioners initially used these as ilioinguinal, iliohypogastric, rectus sheath blocks, and in the early 21st century, transversus abdominis plane (TAP) blocks. A recent variation of the TAP block is known as the quadratus lumborum block (QLB).

The QL block effectiveness is believed to result from the spread of Local Anesthetic cranially from the lumbar deposition into the thoracic paravertebral space (TPVS). So, the QLB seems to relieve somatic and visceral pains.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65 years.
* Both sexes.
* American Society of Anesthesiology (ASA) physical status II-III.
* Body mass index (BMI): (20- 40) kg/m2.
* Type of surgery: midline incision for unilateral open nephrectomy.

Exclusion Criteria:

* Patient refusal.
* Age <18 years or >65 years
* BMI <20 kg/m2 and > 40 kg/m2
* Known sensitivity or contraindication to drugs used in the study
* Contraindication to regional anesthesia, e.g. local infection at the introduction site, pre-existing peripheral neuropathies and coagulopathy.
* Physical status ASA IV
* Patients on chronic analgesic therapy (daily morphine ≥30 mg or equivalent dose of other opioids or tramadol or any medication for neuropathic pain)
* Patients with a history of drug abuse
* Patients with neuropsychiatric diseases; patients with a history of chronic pain syndromes that may enhance sensitivity to pain, for example, fibromyalgia
* All patients who are going to have severe intra- or post-operative bleeding or will require postoperative mechanical ventilation are also excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2025-12-06 (Estimated); Study Completion 2025-12-06 (Estimated)

PRIMARY OUTCOMES:
Degree of pain | 24 hours postoperatively
  The degree of pain will be assessed using the Visual Analogue Scale (VAS) where 0 (no pain) and 10 (the worst pain). VAS score in each technique at 0, 2, 4, 8, 12, 16, 20 and 24 hours postoperatively

SECONDARY OUTCOMES:
Total amount of morphine consumption | 24 hours postoperatively
  Rescue analgesia will be provided in the form of IV morphine 3 mg boluses if the patient indicates Visual Analogue Scale (VAS) ≥ 4. The total amount of morphine given in 24 hours will be recorded for the two groups. A maximum dose of 0.5 mg/kg/24hours of morphine is allowed.
Total amount of fentanyl consumption | Intraoperatively
  Rescue analgesia of fentanyl 1 μg/kg will be given if the mean arterial blood pressure or heart rate rises above 20% of baseline levels.
Change in heart rate | 24 hours postoperatively
  Change in heart rate will be recorded intraoperatively at 5-minute intervals and record the average of each three successive readings, then at 0, 4, 8, 12, 16, 20 and 24 hours postoperatively.
Change in mean arterial blood pressure | 24 hours postoperatively
  Change in mean arterial blood pressure will be recorded intraoperatively at 5-minute intervals and record the average of each three successive readings, then at 0, 4, 8, 12, 16, 20 and 24 hours postoperatively.
Incidence of postoperative nausea and vomiting | 24 hours postoperatively
  Incidence of postoperative nausea and vomiting will be recorded.
Time of first rescue analgesia | 24 hours postoperatively
  Time of first rescue analgesia will be recorded from the end of surgery till first dose of morphine administrated.
Incidence of complications related to block | 24 hours postoperatively
  Incidence of complications related to block such as local anesthetic systemic toxicity and arterial puncture will be recorded.
Incidence of morphine related complications | 24 hours postoperatively
  Incidence of morphine-related complications such as respiratory depression, urine retention or pruritis will be recorded.
Degree of patient satisfaction | 24 hours postoperatively
  The patient will be classified in this group to be satisfied or not.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.